CLINICAL TRIAL: NCT05610189
Title: A Phase 1, Randomized, Multiple-dose, Crossover Trial in Participants With Parkinson's Disease to Evaluate the Clinical Bioequivalence Between Tavapadon Tablets
Brief Title: Multiple-dose Trial to Determine the Clinical Bioequivalence Between Tavapadon Tablets in Participants With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVL-751-1006
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases; Dopamine Agonist; Dopamine Therapy
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Tavapadon 1x15 mg Followed by 3x5 mg (Experimental): Participants will receive tavapadon 1x15 mg tablet, orally, once daily (QD) from Day 15 to 21.
  Participants will receive tavapadon 3x5 mg tablets, orally, QD from Day 22 to 28.
  Interventions: Drug: Tavapadon
- Cohort 2: Tavapadon 3x5 mg Followed by 1x15 mg (Experimental): Participants will receive tavapadon 3x5 mg tablets, orally, QD from Day 15 to 21.
  Participants will receive tavapadon 1x15 mg tablet, orally, QD from Day 22 to 28.
  Interventions: Drug: Tavapadon

INTERVENTIONS:
Drug: Tavapadon — Oral tablets
  Other Names: CVL-751; PF-06649751

SUMMARY:
The primary purpose of the study is to evaluate the bioequivalence (BE) of tavapadon 15 milligram (mg) tablet to 3x5 mg tablets in participants with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index of 17.5 to 38.0 kilograms per square meter (kg/m^2), inclusive, and total body weight >50 kg (110 pounds [lb]) at Screening.
2. Participants with a diagnosis of Parkinson's disease (PD) that is consistent with the United Kingdom (UK) Parkinson's Disease Society Brain Bank diagnostic criteria.
3. Must be modified Hoehn & Yahr Stage I-III inclusive.
4. Must be on a stable dose of L-Dopa of at least 300 mg daily in conjunction with a dopa-decarboxylase inhibitor (e.g., L-Dopa/carbidopa, L Dopa/carbidopa/entacapone or L-Dopa/benserazide) administered at least 3 times per day for at least 2 weeks prior to the Day 1 Visit.

Exclusion Criteria:

1. Participants with a history or clinical features consistent with essential tremor, atypical or secondary parkinsonian syndrome (including, but not limited to, progressive supranuclear palsy, multiple system atrophy, cortico-basal degeneration, or drug-induced or poststroke parkinsonism).
2. Participants with a history of psychosis or hallucinations within the previous 12 months.
3. Participants with epilepsy, or history of epilepsy, or conditions that lower seizure threshold, seizures of any etiology (including substance or drug withdrawal), or who have increased risk of seizures as evidenced by history of electroencephalogram with epileptiform activity are excluded. Participants with a history of febrile seizures only are allowed with medical monitor approval.
4. History of substance or alcohol-use disorder (excluding nicotine; Diagnostic and Statistical Manual of Mental Disorders, 5th edition criteria) within 2 years prior to signing the informed consent form (ICF).
5. Participants who answer "Yes" on the C-SSRS Suicidal Ideation Item 4 (Active Suicidal Ideation with Some Intent to Act, Without Specific Plan) and whose most recent episode meeting criteria for this C-SSRS Item 4 occurred within the last 6 months, OR Participants who answer "Yes" on the C-SSRS Suicidal Ideation Item 5 (Active Suicidal Ideation with Specific Plan and Intent) and whose most recent episode meeting criteria for this C-SSRS Item 5 occurred within the last 6 months OR Participants who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) and whose most recent episode meeting criteria for any of these 5 C-SSRS Suicidal Behavior Items occurred within the last 2 years, OR Participants who, in the opinion of the investigator, present a serious risk of suicide.
6. Participants who have attempted suicide in the past.
7. Positive result for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody with detectable viral ribonucleic acid (RNA) levels at Screening.
8. Have been diagnosed with symptomatic coronavirus disease (COVID-19) or test positive (i.e., using polymerase chain reaction [PCR] or rapid antigen test) for COVID-19 within 30 days prior to signing the ICF.
9. Participants taking strong or moderate cytochrome P450 family 3 subfamily A member 4 (CYP3A4) inducers or inhibitors or who would be likely to require concomitant therapy with CYP3A4 inducers or inhibitors during the trial.

NOTE: Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 28
Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUCτ) of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 28

SECONDARY OUTCOMES:
Minimum Steady-state Plasma Concentration (Cmin,ss) of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 28
Average Steady-state Plasma Concentration (Cavg,ss) of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 28
Trough Concentration (Ctrough) of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 28
Time of Maximum Observed Concentration (Tmax) of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 28
Degree of Fluctuation [(Cmax - Cmin)/Cavg,ss] of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 28
Peak-to-Trough Ratio (PTR) of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 28
Swing [(Cmax - Cmin)/Cmin,ss] of Tavapadon | Pre-dose and at multiple timepoints post-dose up to Day 28
Apparent Clearance of Tavapadon From Plasma (CL/F) | Pre-dose and at multiple timepoints post-dose up to Day 28
Number of Participants With Adverse Events (AEs) and AEs by Severity | Up to Day 36
Number of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Values | Up to Day 29
Number of Participants With Clinically Significant Changes in Vital Sign Values | Up to Day 29
Number of Participants With Clinically Significant Changes in Clinical Laboratory Assessments | Up to Day 29
Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results | Up to Day 29
Changes in Suicidality Assessed Using the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Day 29
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Los Alamitos, California, Los Alamitos, California
  - Hollywood, Florida, Hollywood, Florida
  - Orlando, Florida, Orlando, Florida
  - South Miami, Florida, South Miami, Florida
  - Decatur, Georgia, Decatur, Georgia
  - Farmington Hills, Michigan, Farmington Hills, Michigan

IPD SHARING:
Plan to Share IPD: No